CLINICAL TRIAL: NCT01367769
Title: Evaluation of Perivascular Venous Vascularization and Inflammation by Contrast-enhanced Ultrasound (CEUS) in Patients With Acute Deep Vein Thrombosis and Superficial Thrombophlebitis - a Pilot Study
Brief Title: Venous Vascularization and Inflammation on Contrast-enhanced Ultrasound (CEUS) in Patients With Thrombosis
Status: Terminated | Type: Observational
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: DMS2154
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Thrombosis
Keywords: Deep vein thrombosis; superficial thrombophlebitis; contrast ultrasound
MeSH Terms: conditions — Thrombosis; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators will also determine level of inflammatory markers as the cytokines interleukin-6 (IL-6), interleukin-8 (IL-8), monocyte chemoattractant-1 (MCP-1), Vascular cellular adhesion molecule-1 (VCAM-1), von Willebrand factor (vWF) and C-reactive protein (CRP) at each visit (baseline, 2 weeks, and 3 months).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thrombosis: Patients with acute, idiopathic or provoked, unilateral proximal DVT (involving the popliteal vein or further proximal veins) and SVT of the lower-extremity detected with duplex ultrasound.
  Age and sex matched controls (volunteers)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There will be no intervention in this study.

SUMMARY:
Background:

Contrast-enhanced ultrasound (CEUS) visualization of the adventitial vasa vasorum. Late phase CEUS detect inflammation by visualizing microbubbles phagocytosed by monocytes. The inflammatory process of the vessel wall associated with perivascular angiogenesis at the time of deep venous thrombosis (DVT) and superficial vein thrombophlebitis (SVT) may important in the development of post-thrombotic syndrome (PTS). Therefore the investigators will test the value of CEUS to detect venous perivascular vascularization and inflammation in patients with acute DVT or SVT.

Aims:

To determine the presence and degree of venous perivascular vascularization and inflammation assessed with CEUS in patients with acute DVT or SVT, and compare this to controls without thrombosis.

Expected results:

The investigators hypothesize that venous perivascular vascularization and inflammation assessed by contrast agent enhancement can be quantified and will be significantly more pronounced in the perivascular tissue of the thrombotic vein than in the non affected vein and in controls, and will correlate with level of inflammatory markers and leg volume.

Significance:

These results would provide new information on the pathophysiological concept of thrombosis and thrombus resolution. It might help to better understand the pathophysiologic mechanisms that promote the development of chronic venous insufficiency and PTS.

DETAILED DESCRIPTION:
Background:

Contrast-enhanced ultrasound (CEUS) provides direct in-vivo visualization of the adventitial vasa vasorum using the fact that contrast agents microspheres are ideal intravascular tracers, thus, permitting a non-invasive assessment of the dynamic spatial and temporal heterogeneity of the microvasculature. Moreover, late phase CEUS has shown to detect inflammation by visualizing untargeted microbubbles phagocytosed by monocytes. The inflammatory process of the vessel wall and surrounding tissue associated with perivascular angiogenesis at the time of deep venous thrombosis (DVT) and superficial vein thrombophlebitis (SVT) may promote destruction of venous valves, valvular reflux and subsequent development of post-thrombotic syndrome (PTS). Therefore, in this study, the investigators will test the value of CEUS to detect venous perivascular vascularization and inflammation in patients with acute DVT or SVT.

Aims:

To determine the presence and degree of venous perivascular vascularization and inflammation assessed with CEUS in patients with acute DVT or SVT, and compare this to controls without thrombosis.

Patients and Methods:

20 patients with first unilateral proximal DVT and 10 patients with SVT of the lower-extremity will be included in this study. As control, 10 volunteers without DVT or SVT, and without history of thromboembolism, will be recruited. Diagnosis of DVT and SVT will be performed using standard compression and duplex ultrasound using a Philips (Bothel, WA) ultrasound scanner (iU22) equipped with a linear array L9-4 megahertz (MHz) probe. For CEUS imaging 2.5ml of SonoVueTM (Bracco spa, Milan, Italy) will be injected as an intravenous bolus into an antecubital vein. The thrombotic popliteal vein and the normal popliteal vein at the contralateral side or the thrombotic superficial vein and the normal superficial vein at the contralateral side will be evaluated using a standardized cross-sectional view. Similarly the normal popliteal vein and the superficial vein in a control group will be evaluated. Perivascular contrast-enhancement will be determined with visual interpretation (absent, moderate, abundant) and with quantitative analysis using a dedicated QLAB software (Philips; Bothel, WA) to quantify video intensity within the first minute after bolus contrast injection (perivascular vascularization) and at 6 minutes following the bolus contrast injection (inflammation). Visual based and quantitative analysis of perivascular contrast-enhancement in DVT or SVT will be compared to the contrast-enhancement at the non affected contralateral side and to results of the control group. CEUS imaging with quantification of perivascular contrast-enhancement will be performed at baseline, 2 weeks, and 3 months after acute thrombosis or initial investigation in controls. Additionally, at each visit, measurement of inflammatory markers (MCP-1, IL-6, IL-8, VCAM-1, vWF, and CRP), as well as quantitative measurement of leg volume using an automated 3D image system (Bauerfeind®, Zeulenroda-Triebes, Germany) will be performed.

Expected results:

The investigators hypothesize that venous perivascular vascularization and inflammation assessed by contrast agent enhancement can be quantified and will be significantly more pronounced in the perivascular tissue of the thrombotic vein than in the non affected vein and in controls, and will correlate with level of inflammatory markers and leg volume. Vascularization and inflammation will decrease during the process of thrombus resolution from baseline to 3 months follow-up.

Significance:

These results would provide new information on the pathophysiological concept of thrombosis and thrombus resolution. It might help to better understand the pathophysiologic mechanisms that promote the development of chronic venous insufficiency and post-thrombotic syndrome. As inflammation with pronounced perivascular vascularization might play an important role in incomplete thrombus clearance, venous outflow obstruction and the development of post-thrombotic syndrome after acute DVT, in the future, our results could lead to novel approaches to interrupt the natural history and prevent post-thrombotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* acute, idiopathic or provoked, unilateral proximal DVT (involving the popliteal vein or further proximal veins)
* SVT (more than 5cm in length on compression ultrasonography) of the lower- extremity
* Age and sex matched controls will be recruited from volunteers after exclusion of DVT or SVT, and without history of thrombosis and pulmonary embolism

Exclusion Criteria:

* History of previous DVT or SVT of the lower-extremity
* History of pulmonary embolism
* Bilateral DVT or SVT
* DVT associated with intravenous drug abuse, surgery of the lower-extremity in the previous 10 days, or sclerotherapy in the previous 30 days
* Follow-up is not considered feasible
* Heart failure (HYHA III or IV)
* Acute coronary syndrome (<7d)
* Severe pulmonal-arterial hypertension (pulmonal arterial pressure >90mmHg)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients with unilateral proximal DVT and 10 patients with SVT of the lower-extremity will be included in this study. As control, 10 volunteers without DVT or SVT, and without history of thromboembolism, will be recruited.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Venous perivascular vascularization and inflammation | At baseline, 2 weeks, and 3 months
  Venous perivascular vascularization and inflammation assessed by contrast-enhanced ultrasound

SECONDARY OUTCOMES:
Inflammatory markers | At baseline, 2 weeks, and 3 months
  Interleukin-6 (IL-6), interleukin-8 (IL-8), monocyte chemoattractant-1 (MCP-1), Vascular cellular adhesion molecule-1 (VCAM-1), von Willebrand factor (vWF) and C-reactive protein (CRP)
Edema of the lower extremity | At baselin, 2 weeks, and 3 months
  Quantitative volume measurement of the legs will be performed using an automated 3D image measurement system (Bauerfeind®, Zeulenroda-Triebes, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Staub, MD, Principal Investigator — Unversity Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Staub D, Partovi S, Schinkel AF, Coll B, Uthoff H, Aschwanden M, Jaeger KA, Feinstein SB. Correlation of carotid artery atherosclerotic lesion echogenicity and severity at standard US with intraplaque neovascularization detected at contrast-enhanced US. Radiology. 2011 Feb;258(2):618-26. doi: 10.1148/radiol.10101008. Epub 2010 Oct 22. PMID 20971776
- [Background] Staub D, Schinkel AF, Coll B, Coli S, van der Steen AF, Reed JD, Krueger C, Thomenius KE, Adam D, Sijbrands EJ, ten Cate FJ, Feinstein SB. Contrast-enhanced ultrasound imaging of the vasa vasorum: from early atherosclerosis to the identification of unstable plaques. JACC Cardiovasc Imaging. 2010 Jul;3(7):761-71. doi: 10.1016/j.jcmg.2010.02.007. PMID 20633855
- [Background] Staub D, Patel MB, Tibrewala A, Ludden D, Johnson M, Espinosa P, Coll B, Jaeger KA, Feinstein SB. Vasa vasorum and plaque neovascularization on contrast-enhanced carotid ultrasound imaging correlates with cardiovascular disease and past cardiovascular events. Stroke. 2010 Jan;41(1):41-7. doi: 10.1161/STROKEAHA.109.560342. Epub 2009 Nov 12. PMID 19910551
- [Background] Owen DR, Shalhoub J, Miller S, Gauthier T, Doryforou O, Davies AH, Leen EL. Inflammation within carotid atherosclerotic plaque: assessment with late-phase contrast-enhanced US. Radiology. 2010 May;255(2):638-44. doi: 10.1148/radiol.10091365. PMID 20413774